CLINICAL TRIAL: NCT03371472
Title: Evaluation of the Usefulness of Imaging Methods and 3D Reconstruction in Percutaneous Closure Procedures of Paravalvular Leak (Clinical Trial).
Brief Title: Evaluation of the Usefulness of Imaging Methods and 3D Reconstruction in Percutaneous Closure Procedures of PVL.
Acronym: VALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Protocol Rev 2.0 (2016-09-26)
Record Dates: First submitted 2017-08-10; First posted 2017-12-13 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: PVL - Paravalvular Leak

STUDY DESIGN:
Intervention Model Description: In a group of patients with PVL there are defined two arms: one where PVL is located in mitral position (10 patients) and the second one where PVL is located in aortic position (10 patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VALE - PVL leak sizing balloon - mitral (Other): Placement and inflation of PVL leak sizing balloon for visualisation and measuring of paravalvular leak located in mitral position - Balton developed investigational balloon
  Interventions: Device: Visualisation and measuring of paravalvular leak.
- VALE - PVL leak sizing balloon - aortic (Other): 'Placement and inflation of PVL leak sizing balloon for visualisation and measuring of paravalvular leak located in aortic position - Balton developed investigational balloon
  Interventions: Device: Visualisation and measuring of paravalvular leak.

INTERVENTIONS:
Device: Visualisation and measuring of paravalvular leak. — Visualisation and measurements of PVL by investigational sizing ballons made by Balton. The balloon is a modification of diameter and length of existing sizing ballons (AcuMark™, AMPLATZER™, Occlutech®).

SUMMARY:
Paravalvular leak (PVL) is a condition that could be treated surgically or by the transcatheter deployment of the occluder devices (plugs).

No PVL-specific occluder device is available on the market. VALE consortium plans to design and validate a new PVL dedicated devices (sizing balloon and occluder) in the context of computer 3D modeling, bench testing, preclinical evaluation and clinical research.

DETAILED DESCRIPTION:
Transcatheter closure of PVL has emerged as a new treatment strategy that can be offered to patients with isolated PVL or to those with a very high risk of repeat surgery. The transcatheter approach involves deployment of occlude devices or coils and adopting either a percutaneous or a transapical approach. Limitation of such approach is the fact that no PVL-dedicated device is available on the market, and either vascular-specific plugs or other types of occluders used commonly for closure of ventricular septal defects or patent ductus arteriosus can be used. Several technical issues can make the procedure challenging.

The primary problem is the localization and track of the canal which can be very difficult to engage and cross with the guidewire. Also the maneuverability of the guide catheter in often enlarged left atrium and the passage of the occluder device through narrow and serpiginous canal between calcified annulus and sewing ring is challenging.

Clearly the limitations of current devices and increasing number of patients with significant PVL warrant the attempts to design and validate new PVL-dedicated devices in the context of computer modeling, bench testing, preclinical evaluation and clinical translation. These devices, as sizing balloon, could significantly simplify and shorten the procedure, decrease the risk of complications and incomplete defect closure as well as optimize cost-effectiveness of the procedure by decreasing number of the occluders.

ELIGIBILITY:
Inclusion Criteria:

* The presence of clinically and haemodynamically significant leakage around the surgically implanted cardiac prosthesis in the mitral or aortic position.
* Heart surgery (heart team) disability after another cardiac surgery.
* Technical feasibility of paravalvular leakage closure according to experienced operator.

Exclusion Criteria:

* Active endocarditis on artificial valve
* Instability of artificial valve
* The amount of cavity that prevents effective closure with an occluder
* A history of acute coronary syndrome in less than 3 months before enrollment
* Confirmed echocardiography of transplatin or transesophageal echocardiography
* Hypersensitivity to contrast media
* Any condition associated with the expected life expectancy of less than 6 months
* Haemorrhagic diathesis
* Significant renal impairment (eGFR <30 mL/min/1.73m2)/chronic kidney disease at >G3 stage
* Pregnancy or lactation
* Under 18 years of age
* Patient unable or unwilling to give an informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with sizing procedure success (efficacy outcome) | During index procedure
  Sizing procedure is defined as effective when all following steps: device introduction into the leakage channel, filling in the leakage channel, obtaining a balloon image in the X-ray recording and removal of the balloon without complications are performed.
Incidence of a combined investigational device safety endpoint (safety outcome) | During index procedure
  Safety of the investigational device defined as the occurrence/frequency of locking, fragmentation of the dimensioning balloon, enlargement of the leakage channel, locking of the mechanical prosthesis disks.
  Failure to use the investigational device defined as: locking of the dimensional balloon in site, fragmentation of the dimensional balloon, enlargement of the leakage channel dimension directly related to the application of the dimensional balloon, locking of the mechanical prosthesis disks.
  The failure will be assessed per investigational device and accounted for if at least one of four described events occur. Moreover, the frequency of each event will be additionally assessed and presented in per investigational device analysis.

SECONDARY OUTCOMES:
Frequency of major undesirable cardiovascular events | 30 days observation
  MACCE defined as: cardiac and non-cardiac death, stroke, TIA, myocardial infarction
Frequency and severity of hemorrhagic complications | 30 days observation
  The hemorrhagic complications rated using BARC scale during 30 days follow up
Size of paravalvular leakage after procedure | During index procedure
  Evaluated in transesophageal echocardiography
Comparison of the size of the paravalvular leakage channel illustrated by a dimensional balloon obtained using 3D-TEE and computerized tomography echocardiography | During index procedure
  Comparison of the measurements by sizing balloon to TEE and CT.
Total radiation dose. | During index procedure
  The amount of total radiation dose during index procedure.
Total radiation time. | During index procedure
  The total radiation time of the index procedure.
Duration of the dimensional procedure. | During index procedure
  The duration of the dimensional procedure during index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Wojakowski, Prof., Principal Investigator — III Oddział Kardiologii, Samodzielny Publiczny Szpital Kliniczny nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach, Górnośląskie Centrum Medyczne im. prof. Leszka Gieca
Locations (2):
- Poland (2):
  - II Oddział Kliniczny Kardiologii i Interwencji Sercowo-Naczyniowych, Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - III Oddział Kardiologii, Samodzielny Publiczny Szpital Kliniczny nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach, Górnośląskie Centrum Medyczne im. prof. Leszka Gieca, Katowice, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing data policy is currently restricted under grant consortium agreement and pending GDPR implementation in Europe.

REFERENCES:
- [Background] Smolka G., Wojakowski W., Ochała A., Roleder T., Gąsior Z. Diagnosis and percutaneous treatment of paravalvular leaks; Post Kardiol Interw 2011; 7, 1 (23): 56-60
- [Background] Scognamiglio G, Santoro G, Fusco F, Russo MG, Sarubbi B. Percutaneous treatment of multi-valvular paraprosthetic leaks in a "fragile" heart. Int J Cardiol. 2016 Nov 1;222:790-791. doi: 10.1016/j.ijcard.2016.07.283. Epub 2016 Aug 2. No abstract available. PMID 27521562
- [Background] Murakami T, Fujii H, Sakaguchi M, Takahashi Y, Suehiro Y, Nishimura S, Sakon Y, Yasumizu D, Sohgawa E, Shibata T. Intravascular ultrasound for transcatheter paravalvular leak closure. Gen Thorac Cardiovasc Surg. 2017 Aug;65(8):466-469. doi: 10.1007/s11748-016-0700-x. Epub 2016 Aug 8. PMID 27501692
- [Background] Giacchi G, Freixa X, Hernandez-Enriquez M, Sanchis L, Azqueta M, Brugaletta S, Martin-Yuste V, Masotti M, Sabate M. Minimally Invasive Transradial Percutaneous Closure of Aortic Paravalvular Leaks: Following the Steps of Percutaneous Coronary Intervention. Can J Cardiol. 2016 Dec;32(12):1575.e17-1575.e19. doi: 10.1016/j.cjca.2016.03.013. Epub 2016 Apr 1. PMID 27378589
- [Background] Smolka G, Pysz P, Kozlowski M, Jasinski M, Gocol R, Roleder T, Kargul A, Ochala A, Wojakowski W. Transcatheter closure of paravalvular leaks using a paravalvular leak device - a prospective Polish registry. Postepy Kardiol Interwencyjnej. 2016;12(2):128-34. doi: 10.5114/aic.2016.59363. Epub 2016 May 11. PMID 27279872
- [Background] Cruz-Gonzalez I, Rama-Merchan JC, Calvert PA, Rodriguez-Collado J, Barreiro-Perez M, Martin-Moreiras J, Diego-Nieto A, Hildick-Smith D, Sanchez PL. Percutaneous Closure of Paravalvular Leaks: A Systematic Review. J Interv Cardiol. 2016 Aug;29(4):382-92. doi: 10.1111/joic.12295. Epub 2016 May 31. PMID 27242018
- [Background] Taramasso M, Maisano F, Pozzoli A, Alfieri O, Meier B, Nietlispach F. Catheter-based treatment of paravalvular leaks. EuroIntervention. 2016 May 17;12 Suppl X:X55-X60. doi: 10.4244/EIJV12SXA11. PMID 27174113
- [Background] Hilling-Smith R, Chong A, Cox S. Mitral paravalvular leak closure by antegrade percutaneous approach using amplatzer PFO closure device. Catheter Cardiovasc Interv. 2017 Aug 1;90(2):E62-E67. doi: 10.1002/ccd.26417. Epub 2016 Apr 16. PMID 27084789
- [Background] Abdelghani M, Soliman OI, Schultz C, Vahanian A, Serruys PW. Adjudicating paravalvular leaks of transcatheter aortic valves: a critical appraisal. Eur Heart J. 2016 Sep 7;37(34):2627-44. doi: 10.1093/eurheartj/ehw115. Epub 2016 Apr 13. PMID 27075871